CLINICAL TRIAL: NCT03130179
Title: A Single-dose, Two-period, Crossover, Randomized, Fasting, Open-label, Bioequivalence Study Between Nicorette Strongmint Lozenge 4 mg and Niquitin Minimint Lozenge 4 mg in Adult Healthy Smokers Motivated to Quit.
Brief Title: A Bioequivalence Study Between Two Nicotine Replacement Therapies in Adult Healthy Smokers Motivated to Quit.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: McNeil AB (Industry)
Responsible Party: Sponsor
Organization: Johnson & Johnson Consumer and Personal Products Worldwide (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: CO-141210150531-SCCT
Record Dates: First submitted 2017-03-29; First posted 2017-04-26 (Actual); Last update posted 2018-07-27 (Actual); Status verified 2018-06

CONDITIONS: Tobacco Dependence
Keywords: Bioequivalence
MeSH Terms: conditions — Tobacco Use Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nicorette Strongmint lozenge 4mg (Experimental): A single dose of one nicotine 4 mg lozenge will be administrated orally to slowly dissolve in the mouth for nicotine absorption via the buccal mucosa.
  Interventions: Drug: Nicorette Strongmint lozenge 4 mg
- Niquitin Minimint lozenge 4mg (Active Comparator): A single dose of one nicotine 4mg lozenge will be administrated orally to slowly dissolve in the mouth for nicotine absorption via the buccal mucosa.
  Interventions: Drug: Niquitin MiniMint lozenge 4 mg

INTERVENTIONS:
Drug: Nicorette Strongmint lozenge 4 mg — A single dose of one Nicorette lozenge 4mg lozenge administrated orally to slowly dissolve in the mouth.
  Other Names: Nicorette lozenge 4 mg
  Arms: Nicorette Strongmint lozenge 4mg
Drug: Niquitin MiniMint lozenge 4 mg — A single dose of one Niquitin Minimint lozenge 4mg administrated orally to slowly dissolve in the mouth.
  Other Names: Niquitin lozenge 4 mg
  Arms: Niquitin Minimint lozenge 4mg

SUMMARY:
This is a research study to verify the same effectiveness and safety profile for the test product, Nicorette Strongmint lozenge, as for an already approved product, NiQuitin® Minimint lozenge (reference product), in a standardized mode. This verification is done in a so-called bioequivalence study, which means that the same amount of the same active substance (nicotine), in the same dosage form, for the same route of administration, and meeting the same or comparable standards is performed.

During the study visits, blood samples will be drawn to measure the level of the substance in the blood to verify that the two products are comparable. Tolerability of the treatments will be evaluated based on reported and observed adverse events.

DETAILED DESCRIPTION:
This is a single-dose, two-period crossover, randomized, fasting, open-label, bioequivalence study.

244 male and female volunteers with a smoking history of minimum 3 months and aged between 18 and 45 years, inclusive, and motivated to quit will be included. The treatment administration order will be randomized with an equal number of subjects in each treatment sequence.

Single doses of 4 mg Nicorette Strongmint Lozenge (i.e. test product) and 4 mg NiQuitin® Minimint Lozenge (i.e. reference product) will be administered in a standardized mode, on two separate treatment visits. A washout period of minimum 48 hours will separate the treatment administrations.

An abstinence period of 12 hours including an overnight stay at the clinic is required at both treatment occasions.

Blood for pharmacokinetic analyses will be drawn pre-dose (i.e. within 5 minutes before drug administration) and at 10, 15, 20, 30, 40, 50, and 60 minutes, as well as 1.25, 1.5, 2, 3, 4, 6, 8, 10, and 12 hours after start of drug administration. Thus, 17 samples will be collected per treatment visit.

Subjects will be monitored to capture any adverse events that may occur.

ELIGIBILITY:
Inclusion Criteria:

1. Male and/or female subjects 18 to 45 years of age, inclusive, and being verified "Healthy". ("Healthy" is defined as absence of any diseases or abnormalities on the basis of physical examination, standard clinical laboratory and instrumental examinations performed at the screening visit).
2. Smoking at least 10 tobacco cigarettes daily for at least three months preceding inclusion and presence of motivation to quit smoking.
3. Subjects with a Body Mass Index (BMI) between 18.5 to 30 kg/m2, inclusive, and a body weight >50 kg.
4. Females of childbearing potential must have a negative urine pregnancy test at the screening visit.
5. Male or non-pregnant, non-lactating female agree to the contraceptive requirements (including male's and female partner's use of a highly effective methods of birth control for at least 3 months before the study, during the study and for 30 days after the last dose of study drug) as outlined in Section 10.7
6. Has a personally signed and dated informed consent document before participating in any study-specific procedures, indicating that the subject has been informed of all pertinent aspects of the study; and
7. Is able to comprehend the requirements of the study (based upon clinical site personnel's assessment), and is willing and able to comply with scheduled visits,treatment plan, laboratory tests, and other study procedures specified in the protocol.

Exclusion Criteria:

1. Deviations from normal ranges as a result of standard clinical laboratory and instrumental examinations including ECG, performed at the screening visit.
2. Use of vitamins, herbal supplements and medicinal plants (e.g. garlic) within 7 days before the first dose of study medication. Use of products containing St. John's wort [Hypericum perforatum] 30 days prior to the study start.
3. Intake of medications having a significant impact on hemodynamics, hepatic function etc. (e.g. [but not limited to] barbiturates, omeprazole cimetidine).
4. Subjects who will not abstain from using nicotine-containing products (besides treatments specified in this protocol) and smoking from 12 hours before planned treatment intake and throughout each visit.
5. Is hypersensitive, intolerant, or experienced an allergic reaction to the active ingredient(s) or excipients of drug products that will be used in the study or has severe allergy (e.g. anaphylaxis, angioedema) in the past.
6. Females with a positive pregnancy test and/or are breast-feeding.
7. Females, currently using hormonal contraceptives, (including use less than 2 weeks prior to enrollment)
8. Males with a pregnant spouse or partner or males who are not willing to prevent conception in a spouse or partner.
9. Has a positive test for human immunodeficiency virus (HIV) 1 and 2 antibodies, hepatitis B surface antigen (HBsAg), or hepatitis C antibodies (anti-HCV) or syphilis (RW).
10. Has a positive test for psychoactive and narcotic substances, psychoactive drugs at screening and/or at any admission to the clinical center or has drugs abuse in the past.
11. Consumes alcohol regularly in excess of the following: >10 units per week (1 unit of alcohol is equivalent to ½ liter of beer, 200 ml wine or 50 ml of vodka) or presence of information on alcoholism in medical history. The subject must also abstain from alcohol consumption within 48 hours prior to the screening visit and have a negative respiratory alcohol test at the screening visit and/or at any admission clinical center (breathalyzer).
12. Use of xanthine products within 48 hours prior to the first dose of the investigational product.
13. Ingestion of food or beverages containing grapefruit, Chinese grapefruit (pomelo) or Seville oranges (including marmalade) within 10 days prior to the first dose of the investigational product and inability to stop these products taking during the study.
14. Abuse of caffeine products exceeding 500mg caffeine daily (5 cups of coffee) and the ability to abstain from caffeine products at least 48 hours before the first dose of investigational product intake and prior to prior to collection of the last blood sample in each period of the study.
15. Renal or hepatic impairment.
16. Has a history of gastrointestinal surgery other than appendectomy, ulcers or any other lesions in the mouth.
17. Erosive and ulcerative lesions of oral mucosa, xerostomia, including a history of these diseases, jaw trauma and surgery.
18. Heart rate < 60 or > 80 per minute at rest, or systolic blood pressure <100 or >130 mm Hg, or diastolic blood pressure < 70 or > 90 mm Hg.
19. Acute infections within 4 weeks prior to the study.
20. Treatment with an investigational drug within 3 months preceding the first dose of study treatment.
21. Donation of ≥450mL blood or plasma, or loss of ≥500mL of blood 3 months prior to the first of investigational product intake.
22. Preplanned surgery or procedures during the study period, if this may interfere with the conduct of the study.
23. Inability to give written informed consent or comply with the protocol requirements.
24. Probability to refuse to comply with the protocol requirements, instructions and restrictions; for example, unwillingness to cooperate, inability to return to the clinical center for follow-up visits and the probability of incomplete participation in the clinical trial.
25. Participation in clinical trials less than 3 months prior to the study.
26. Relationship to persons involved directly with the conduct of the study (i.e., principal investigator; sub investigators; study coordinators; other study personnel; employees or contractors of the Sponsor or Johnson & Johnson subsidiaries; and the families of each).

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 244 (Actual)
Dates: Start 2017-03-20 (Actual); Primary Completion 2017-06-19 (Actual); Study Completion 2017-06-29 (Actual)

PRIMARY OUTCOMES:
Peak Plasma Concentration (Cmax) of nicotine | At baseline, 10, 15, 20, 30, 40, 50 and 60 minutes, 1.25, 1.5, 2, 3, 4, 6, 8, 10 and 12 hours after start of drug administration.
  The maximum observed plasma concentration (Cmax)
The time at which the maximum nicotine concentration (Cmax) occurs (Tmax) | At baseline, 10, 15, 20, 30, 40, 50 and 60 minutes, 1.25, 1.5, 2, 3, 4, 6, 8, 10 and 12 hours after start of drug administration.
  Tmax is defined as the time point at which the maximum nicotine concentration (Cmax) occurs
Area under the plasma concentration versus time curve (AUCt) from start of nicotine administration until the last measurable concentration. | At baseline, 10, 15, 20, 30, 40, 50 and 60 minutes, 1.25, 1.5, 2, 3, 4, 6, 8, 10 and 12 hours after start of drug administration.
  AUCt is defines as area under the plasma concentration versus time curves from start of drug administration until the last measureable concentration.
Area under the plasma concentration versus time curve (AUC∞) of nicotine | At baseline, 10, 15, 20, 30, 40, 50 and 60 minutes, 1.25, 1.5, 2, 3, 4, 6, 8, 10 and 12 hours after start of drug administration.
  AUC∞ is defined as area under the plasma concentration versus time curves from start of drug administration until the nicotine plasma concentration is negligible (infinity).
The extrapolated part of area under the plasma concentration versus time curve (AUC∞) of nicotine. | Extrapolation from 12 hours after start of drug administration until infinity.
  The area under the plasma concentration versus time curves from start of drug administration until infinity.
Determination of the terminal elimination rate constant (lambda_z) for nicotine. | At baseline, 10, 15, 20, 30, 40, 50 and 60 minutes, 1.25, 1.5, 2, 3, 4, 6, 8, 10 and 12 hours after start of drug administration.
  The rate at which the drug is removed from the body system.
The plasma half-life (t1/2) of nicotine. | At baseline, 10, 15, 20, 30, 40, 50 and 60 minutes, 1.25, 1.5, 2, 3, 4, 6, 8, 10 and 12 hours after start of drug administration.
  The time taken for the nicotine plasma concentration to fall to half its original value.

SECONDARY OUTCOMES:
Percentage of Subjects with Treatment-Emergent Adverse Events after single-dose administration of Nicorette Strongmint Lozenge 4mg or NiQuitin Minimint Lozenge 4mg. | From first dose received up to 3.5 weeks + 30 days follow up after study completion for any unresolved adverse events.
  Frequency (%) of subjects experiencing treatment-emergent adverse events by treatment, system organ class and preferred term.
Percentage of Subjects with Treatment-Emergent Adverse Events after single-dose administration of Nicorette Strongmint Lozenge 4mg or NiQuitin Minimint Lozenge 4mg - By Worst-Case Severity. | From first dose received up to 3.5 weeks + 30 days follow up after study completion for any unresolved adverse events.
  Frequency (%) of subjects experiencing treatment-emergent adverse events by treatment, system organ class, preferred term and severity.
Percentage of Subjects with common treatment-emergent adverse events (AEs) after single-dose administration of Nicorette Strongmint Lozenge 4mg or NiQuitin Minimint Lozenge 4mg. | From first dose received up to 3.5 weeks + 30 days follow up after study completion for any unresolved adverse events.
  Percentage (%) of subjects with commonly reported treatment-emergent adverse events by system organ class and preferred term.
Percentage of Subjects with treatment-related adverse events (AEs) after single-dose administration of Nicorette Strongmint Lozenge 4mg or NiQuitin Minimint Lozenge 4mg. | From first dose received up to 3.5 weeks + 30 days follow up after study completion for any unresolved adverse events.
  Percentage (%) of subjects experiencing treatment-related adverse events by treatment, system organ class and preferred term.
Percentage of Subjects with treatment-related adverse events (AEs) after single-dose administration of Nicorette Strongmint Lozenge 4mg or NiQuitin Minimint Lozenge 4mg - By Worst-Case Severity. | From first dose received up to 3.5 weeks + 30 days follow up after study completion for any unresolved adverse events.
  Percentage (%) of subjects experiencing treatment-related adverse events by treatment, system organ class, preferred term and severity.
Percentage of Subjects with treatment-emergent serious adverse events (SAEs). | From first dose received up to 3.5 weeks + 30 days follow up after study completion.
  Percentage (%) of subjects experiencing treatment-emergent serious adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Elena P Mazygula, MD, Principal Investigator — "Scientific and Clinical Center of JSC "RZD"
Locations (1):
- "Scientific and Clinical Center of JSC "RZD", Moscow, Russia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: CSR Synopsis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_7051&studyid=12386&filename=Final%20Approved%20CSR%20Synopsis_marked%20for%20redaction_Redacted.pdf